CLINICAL TRIAL: NCT01152957
Title: Miami Healthy Heart Initiative (MHHI) a Randomized Study of Behavioral Risk Factors for Cardiovascular Disease in Latino and Hispanic Patients With Poorly Controlled Diabetes
Brief Title: Miami Healthy Heart Initiative a Behavioral Study on Cardiovascular Risk Factors
Acronym: MHHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Olveen Carrasquillo, Chief, Division of General Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20090751; 7R01HL083857-02 (NIH)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Diabetes; Heart Disease; Hypertension
Keywords: diabetes; cardiovascular; chronic; Community Health Workers; behavioral; social; diet; exercise; patient; cholesterol; A1C; blood pressure
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Hypertension; Bronchiolitis Obliterans Syndrome; Behavior; Motor Activity

STUDY DESIGN:
Masking Description: single blinded
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Community Health Worker Model (Experimental): Care, Attention, Resources, Information, Nutrition and Optimism Project (CARIÑO Project) will provide outreach support services to patients with poorly controlled diabetes, such as health education, lifestyle changes, home visits, follow-up phone calls, support groups, one on one counseling and coaching, and assistance with resource referrals.
  Interventions: Behavioral: CARIÑO Project
- Enhanced Usual Care (Active Comparator): Usual Care and mailing of 4 health education brochures over the year.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: CARIÑO Project — Care Attention Resources Information Nutrition & Optimism Project (CARIÑO) is a CHW intervention that will involve 4 or more (as required) home visits, 10 group sessions, and 10 follow-up phone calls per subject over a 12-month period. The primary outcome is lower HgA1C levels. The secondary outcomes are to lower LDL levels, and systolic and diastolic blood pressure, medication adherence and improved diet and exercise. CARIÑO Project will provide outreach support services to patients with poorly controlled diabetes, such as health education, lifestyle changes, home visits, follow-up phone calls, support groups, one on one counseling and coaching, and assistance with resource referrals.
  Arms: Community Health Worker Model
Behavioral: Enhanced Usual Care — Usual care plus 4 health education brochures
  Arms: Enhanced Usual Care

SUMMARY:
A study to examine the effectiveness of a multilevel Community Health Workers intervention as an adjunct to routine primary care in reducing CVD risk factors among diabetic Latinos in Miami.

DETAILED DESCRIPTION:
Disparities in the epidemiology of cardiovascular disease (CVD) risk factors among Latinos have been extensively described; however, traditional medical models of CVD risk reduction have not been very effective in Latinos. One promising strategy is the use of community-based community health workers (CHWs). CHWs have long been used in Latin-America as an integral part of their health care delivery system. Further, preliminary data from our prior pilot diabetes self-management CHW program have shown improvements in lipids. However, because of a lack of effectiveness data from studies using rigorous experimental designs, the adoption of the CHW model has been quite limited both locally and nationally. In MHHI, our goal is to examine the effectiveness of a CHW intervention in CVD risk reduction among Latinos.

The investigators propose to examine the effectiveness of a multilevel CHW intervention as an adjunct to routine primary care in reducing CVD risk factors among diabetic Latinos Miami. The UM Jay Weiss Center which has substantial experience in Community Health Worker Program will take the lead role in the development and implementation intervention of the CHW program.

The study design is a randomized controlled trial (RCT) of 300 Latino patients ages 35-70 with poorly controlled diabetes (AIC >=8.0) followed at the Ambulatory Care Clinic (ACC) of Jackson Memorial Hospital (JMH).

Primary Objective: To determine if the CHW intervention results in lowering of CVD risk factors including blood pressure, LDL cholesterol, and diabetes control (AIC) as measured by the Total Framingham Risk Score (FRS).

Secondary Objectives: To determine if the CHW intervention results in improvements in the following putative mechanisms that may influence the FRS:

1. Medication adherence (measured by validated instruments)
2. Improvements in diet and exercise (as measured by validated instruments);

Hypotheses: Among patients receiving care at the ACC we hypothesize that as compared to those in enhanced usual care, patients randomized to the CHW intervention at 18 months will have:

1. Greater reductions in blood pressure and low density lipoprotein (LDL)
2. Improved glycemic control
3. Greater rates of medication adherence (taking >80% of specified medication doses)
4. Increases in physical activity (kcal/week)
5. Increases in mean number of daily vegetables consumed

The CHW intervention will involve 4 or more (as required) home visits, 10 group sessions, an 10 follow-up phone calls per subject over a 12-month time period. The primary outcome is a HgA1C; secondary outcomes include LDL levels, and systolic and diastolic blood pressure. Baseline and follow-up data on medication adherence, medication intensification, diet and exercise will also be collected.

The control group will continue to receive usual care from their primary care physician. We will enhance the usual care that these patients receive by providing them with three sets of educational materials published by the NIH.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 35-70 years
* Receiving care at ACC clinic (2 visits with a primary care provider in the previous year)
* Living in Miami-Dade county (based on zip codes)
* Had a hemoglobin A1C done within the past year, with the latest value being >=8.0

Exclusion Criteria:

* Patients whose Primary Doctor believes are not appropriate candidates for participation
* Type 1 diabetics (identified by Primary Doctor or those with diabetes diagnosed when under age 25).
* Patients who do not self identify as Hispanic
* Any life-threatening or extreme medical comorbidity
* Having a diabetes diagnosis for less than a year
* Planning to move out of the neighborhood during the next year
* Participation in any other CVD or diabetes intervention study
* Arm circumference of greater than 47 cm (oscillometric cuffs do not give accurate readings)

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Glycemic Control | 12 months.
  A1C

SECONDARY OUTCOMES:
Blood Pressure | 12 months
  SBP
Cholesterol | 12 months
  LDL

CONTACTS AND LOCATIONS:
Overall Officials: Olveen Carrasquillo, MD, MPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Contact PI

REFERENCES:
- [Background] Carrasquillo O, Patberg E, Alonzo Y, Li H, Kenya S. Rationale and design of the Miami Healthy Heart Initiative: a randomized controlled study of a community health worker intervention among Latino patients with poorly controlled diabetes. Int J Gen Med. 2014 Feb 27;7:115-26. doi: 10.2147/IJGM.S56250. eCollection 2014. PMID 24600243
- [Background] Kenya S, Lebron CN, Chang AY, Li H, Alonzo YA, Carrasquillo O. A profile of Latinos with poorly controlled diabetes in South Florida. J Community Hosp Intern Med Perspect. 2015 Apr 1;5(2):26586. doi: 10.3402/jchimp.v5.26586. eCollection 2015. PMID 25846350
- [Background] Lebron CN, Reyes-Arrechea E, Castillo A, Carrasquillo O, Kenya S. Tales from the Miami Healthy Heart Initiative: the experiences of two community health workers. J Health Care Poor Underserved. 2015 May;26(2):453-62. doi: 10.1353/hpu.2015.0033. PMID 25913343
- [Background] Chang A, Kenya S, Ilangovan K, Li H, Koru-Sengul T, Alonzo Y, Carrasquillo O. Is greater acculturation associated with an increased prevalence of cardiovascular risk factors among Latinos in South Florida? Med Care. 2015 May;53(5):417-22. doi: 10.1097/MLR.0000000000000337. PMID 25793266
- [Result] Carrasquillo O, Lebron C, Alonzo Y, Li H, Chang A, Kenya S. Effect of a Community Health Worker Intervention Among Latinos With Poorly Controlled Type 2 Diabetes: The Miami Healthy Heart Initiative Randomized Clinical Trial. JAMA Intern Med. 2017 Jul 1;177(7):948-954. doi: 10.1001/jamainternmed.2017.0926. PMID 28459925
- [Result] Chang A, Patberg E, Cueto V, Li H, Singh B, Kenya S, Alonzo Y, Carrasquillo O. Community Health Workers, Access to Care, and Service Utilization Among Florida Latinos: A Randomized Controlled Trial. Am J Public Health. 2018 Sep;108(9):1249-1251. doi: 10.2105/AJPH.2018.304542. Epub 2018 Jul 19. PMID 30024805